CLINICAL TRIAL: NCT04867330
Title: Induction Chemotherapy of Toripalimab With Docetaxel and Cisplatin Followed by De-escalation of Chemoradiotherapy Density in HPV-related Oropharyngeal Carcinoma in Chinese Populations
Brief Title: Toripalimab Based Induction Chemotherapy Followed by De-escalation Protocols in HPV-related OPSCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, Professor, Fudan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-OR001
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Oropharyngeal Carcinoma; Immune Checkpoint Inhibitor; De-escalation
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- conventional treatment arm (Experimental): Two cycles Toripalimab+docetaxel+cisplatin induction chemotherapy followed by concurrent cisplatin chemoradiotherapy with standard radiation dose (70Gy/35Fx) when responses to induction chemotherapy are less than 50% Partial Response(PR)
  Interventions: Other: Toxicities reduced treatment arm

INTERVENTIONS:
Other: Toxicities reduced treatment arm — Two cycles Toripalimab+docetaxel+cisplatin induction chemotherapy followed by reducing radiation dose(60Gy/30Fx) and omitting concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 50% Partial Response(PR)

SUMMARY:
Human papillomavirus (HPV)-related oropharyngeal carcinoma are exquisitely radiosensitive. Several studies attempted to reduce the toxicities of treatments through reduced-dose radiation and showed promising results, but all data were collected from non-Chinese areas. Like nasopharyngeal carcinoma (NPC), oropharyngeal carcinoma may have different biological behavior and relationship with HPV infection. So the investigators studied whether toxicities reducing treatment with reduced radiation dose and omitted concurrent chemotherapy after good response to induction chemotherapy would maintain survival outcomes while improving tolerability for patients with HPV-positive oropharyngeal carcinoma. Immune checkpoint inhibitors (ICIs) have proved to improve outcomes of head and neck cancers including EBV-related NPC. Oropharyngeal carcinoma was considered to be similar with NPC in terms of immune environment. So we added anti-PD-1 antibody Toripalimab to induction chemotherapy in order to achieve better response rates to receive de-escalation chemoradiotherapy followed.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of squamous cell carcinoma of oropharynx with IHC p16
* positive or PCR HPV16 positive
* T1-2/N1-3M0（except T1N1M0 and single LN<3cm）or T3-4N0-3M0 according to UICC/AJCC 8th staging system
* Age ≥18
* No prior anti-tumor treatment
* Karnofsky Performance Score (KPS)≥70
* Adequate blood supply
* Informed consent obtained

Exclusion Criteria:

* Cannot take contrast-MRI imaging
* Pregnant
* Combined with other malignant tumor (except basal cell carcinoma of skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
PFS PFS | 2 year
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, China